CLINICAL TRIAL: NCT05968963
Title: Electronic Health Mindfulness-based Music Therapy Intervention for Patients Undergoing Allogeneic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230726; 1R61CA263335-01A1 (NIH)
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stem Cell Transplantation; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Music Therapy (MBMT) (Experimental): Participants will be in the MBMT group for 5 months.
  Interventions: Behavioral: Mindfulness-based Music Therapy (MBMT)
- Mindfulness Meditation (MM) (Experimental): Participants will be in the MM group for 5 months.
  Interventions: Behavioral: Mindfulness Meditation (MM)

INTERVENTIONS:
Behavioral: Mindfulness-based Music Therapy (MBMT) — Participants will receive 8 music therapy sessions that will last approximately 60 minutes in length. A Music therapist will conduct the sessions. These sessions will be in person and/or virtual depending on patient status and the time between sessions will vary based on patient response to treatment.
  Arms: Mindfulness-based Music Therapy (MBMT)
Behavioral: Mindfulness Meditation (MM) — Participants will receive 8 mindfulness meditation sessions that will last approximately 60 minutes in length. These sessions will be participant led virtually.
  Arms: Mindfulness Meditation (MM)

SUMMARY:
The goal of this study is to pilot test an Electronic Health Mindfulness-based Music Therapy Intervention (eMBMT) intervention to improve health-related quality of life (HRQoL) and reduce symptom burden of patients undergoing allogeneic stem cell transplantation (allo-SCT).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* have a primary diagnosis of myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or non Hodgkin's Lymphoma (NHL)
* have a treatment plan for an allogeneic hematopoietic stem cell transplant
* Speak English or Spanish

Exclusion Criteria:

* history of severe psychiatric illness (e.g., psychosis, active suicidality, inpatient treatment in the past 12 months)
* severe cognitive impairment (per the short portable mental status questionnaire)
* hearing impairment
* active alcohol or substance dependence within the past six months
* participated in music therapy or mindfulness programs in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Count of Participants Recruited | Baseline (T1)
  Recruitment will be measured by the count of participants successfully recruited and randomized into the study.
Number of Participants Retained | Up to 18 months
  Participant retention will be examined via the number of participants retained in the study.
Mean Number of Intervention Sessions that Participants Completed | Up to 100 days post-transplant
  Participant engagement will be examined via the mean number of intervention sessions completed by participants measured after the 8th (and last) intervention session which is given between 75 and 100 days post-transplant.
Satisfaction Scores as Measured by Weekly Rating Satisfaction Score | Up to 100 days post-transplant
  Scores per item range from 0 to 5. Higher scores indicate more satisfaction.

SECONDARY OUTCOMES:
Change in Health Related Quality of Life Scores as Measures by Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) | Baseline (T1), up to 18 months
  FACT-BMT score range 0-164, with higher scores indicating better quality of life.
Change in Pain as Measured by patient reported outcome measures (PROMIS®) pain scale. | Baseline (T1), up to 18 months
  (PROMIS®) pain scale is scored on a range of 3 to 15 with higher scores indicating higher pain.
Change in Fatigue as Measured by patient reported outcome measures (PROMIS®) Fatigue scale. | Baseline (T1), up to 18 months
  (PROMIS®) Fatigue scale is scored on a range of 8 to 40. Higher scores indicate higher fatigue.
Change in Cognitive Function Scores as Measured by The Repeatable Battery for the Assessment of Neuropsychological Status. | Baseline (T1), up to 18 months
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores range from 40-160 with higher scores indicating better cognitive function.
Change in Sleep Quality Scores as Measured by Pittsburgh Sleep Quality Index | Baseline (T1), up to 18 months
  Pittsburgh Sleep Quality Index score range from 0 to 21. Higher score indicate worse sleep quality.
Number of Days to Engraftment Measured from Infusion to Engraftment. | Up to 18 months
  To measure the number of days to engraftment we will extract from the electronic medical record (EMR) days from infusion to engraftment.
Number of Days of Hospitalization Measured from Admission to Engraftment. | Up to 18 months
  To measure the number of days of hospitalization we will extract from the electronic medical record (EMR) days of hospitalization from admission to engraftment.
Number of Hospital Readmissions after Hospital Discharge | Up to 100 days
  To measure the number of hospital readmissions we will extract from the electronic medical record (EMR) the number of hospital readmissions from hospital discharge.
Number of Infections from Hospital Admission | up to 100 Days Post-Infusion Day
  To measure the number of infections we will extract from the electronic medical record (EMR) the number of infections from hospital admission measure up to 100 days post infusion.
Change in anxiety Scores as Measured with the Generalized anxiety disorder (GAD-7) | Baseline (T1), up to 18 months
  Generalized anxiety disorder (GAD-7) range is 0 to 21; higher score is associated with more severe anxiety.
Changes in Depression Scores as measured with the patient health questionnaire (PHQ-9) | Baseline (T1), up to 18 months
  PHQ-9 (patient health questionnaire) score range is from 0 to 27; higher score is associated with more severe depression.
Change in Cancer-specific Distress Scores as Measured by the Impact of Events Scale-Revised | Baseline (T1), up to 18 months
  Impact of Events Scale-Revised range is 0 to 88; higher score is associated with more effect caused by events.
Change in Serum Cortisol as Measured by ELISA | Baseline (T1), up to 18 months
  Serum cortisol levels are measured via ELISA. Serum Cortisol normal levels morning range: 10-20 mcg/dL ; afternoon range: 3-10 mcg/dL. Any values outside of the range are associated with higher stress and inflammation
Change in Immunocompetence as Measured by Cytokines | Baseline (T1), up to 18 months
  Cytokines levels are measured in pg/mL. Any values outside of the normal range are associated with inflammation
Change in Immunocompetence as Measured by Thymic Function | Baseline (T1), up to 18 months
  Thymic function T-cell receptor excision circles (TRECs) measured by TRECs/microliter.
Change in Immunocompetence as Measured by Regulatory T cells | Baseline (T1), up to 18 months
  Regulatory T cells measured as cells/mm^3

CONTACTS AND LOCATIONS:
Overall Officials: Frank J. Penedo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No